CLINICAL TRIAL: NCT01860118
Title: LRRK2 and Other Novel Exosome Proteins in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Andrew B. West, Associate Professor, University of Alabama at Birmingham
Other Study IDs: X121207003; 1U18NS082132 (NIH)
Record Dates: First submitted 2013-04-19; First posted 2013-05-22 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's Disease: 1) the presence of bradykinesia and either rest tremor or rigidity; 2) asymmetric onset; 3) progressive motor symptoms 4) age at onset 21-99 years.
- Healthy Control: Healthy controls between ages of 21-99 years and a lack of PD in first-degree blood relatives

SUMMARY:
This proposal seeks to 1) determine whether there are biomarkers associated with Parkinson's disease (PD) susceptibility and/or progression in exosome-proteomes derived from PD patients versus controls, and 2) to determine if LRRK2 expression and/or phosphorylation are significantly lowered in the exosomes of individuals treated with the potent LRRK2 kinase inhibitor sunitinib (a multi-kinase inhibitor compound), to establish an assay for on-target effects for future LRRK2 inhibitor clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Parkinson's disease inclusion criteria:

Inclusion criteria will be based on UK Brain Bank criteria for the clinical diagnosis of PD. These require 1) the presence of bradykinesia and either rest tremor or rigidity; 2) asymmetric onset; 3) progressive motor symptoms 4) age at onset 21-99 years.

Control inclusion criteria: ages of between 21-99 years, a lack of PD in first-degree blood relatives, and a lack of positive responses on more than 3 items on the PD Screening Questionnaire.

Exclusion Criteria:

For all subjects:

include atypical features indicative of a Parkinson-Plus disorder (Progressive Supranuclear Palsy (PSP), Multiple System Atrophy (MSA), Corticobasal Degeneration (CBD)) including cerebellar signs, supranuclear gaze palsy, apraxia and other cortical signs, or prominent autonomic failure, neuroleptic treatment at time of onset of parkinsonism, active treatment with a neuroleptic at time of study entry, History of repeated strokes with stepwise progression of parkinsonism, history of repeated head injury, history of definite encephalitis, prominent gait imbalance early in the course (< 5 years), dementia, known severe anemia (hematocrit <30), history of kidney disease and/or current or past glomerular filtration rate (GFR) <60 possibly indicative of kidney disease, or a serious comorbidity that may interfere with participation in the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neurology clinic
Sampling Method: Non-Probability Sample
Enrollment: 601 (Actual)
Dates: Start 2013-01; Primary Completion 2016-06-21 (Actual); Study Completion 2016-06-21 (Actual)

PRIMARY OUTCOMES:
Biomarkers | up to 3 years
  Biomarkers associated with Parkinson's disease (PD) susceptibility and/or progression in exosome-proteomes derived from PD patients versus controls.

SECONDARY OUTCOMES:
LRRK2 expression and/or phosphorylation | up to 3 years
  Determine if LRRK2 expression and/or phosphorylation are significantly lowered in the exosomes of individuals treated with the potent LRRK2 kinase inhibitor sunitinib (a multi-kinase inhibitor compound), to establish an assay for on-target effects for future LRRK2 inhibitor clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew West, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Sparks Center, Birmingham, Alabama, United States